CLINICAL TRIAL: NCT05063630
Title: Intracranial Stenting in Non-acute Symptomatic Ischemic Stroke: an Open-label, Randomised Controlled Trial
Brief Title: Intracranial Stenting in Non-acute Symptomatic Ischemic Stroke
Acronym: INSIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Can Tho Stroke International Services Hospital (Other)
Responsible Party: Principal Investigator, Dr. Cuong Tran Chi, Director - Doctor, Can Tho Stroke International Services Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CanTho S.I.S Hospital
Record Dates: First submitted 2021-09-15; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Intracranial Arteriosclerosis; Ischemic Stroke; Intracranial Arterial Diseases; Arterial Occlusive Diseases
Keywords: Dual antiplatelet therapy; MRI 3 Tesla; WEAVE trial; WOVEN trial
MeSH Terms: conditions — Intracranial Arteriosclerosis; Ischemic Stroke; Intracranial Arterial Diseases; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical treatment plus intracranial stenting (MT plus IS) (Experimental): This group will be both given medical treatment (aspirin 100 mg and clopidogrel 75 mg per day for 90 consecutive days and clopidogrel 75 mg per day thereafter) and performed with intracranial stenting.
  Interventions: Procedure: Medical treatment plus intracranial stenting
- Medical treatment alone (MT) (Active Comparator): This group will be given medical treatment including aspirin 100 mg and clopidogrel 75 mg per day for 90 consecutive days and clopidogrel 75 mg per day thereafter.
  Interventions: Drug: Medical treatment alone

INTERVENTIONS:
Procedure: Medical treatment plus intracranial stenting — This group will be both given medical treatment (aspirin 100 mg and clopidogrel 75 mg per day for 90 consecutive days and clopidogrel 75 mg per day thereafter) and performed with intracranial stenting.
  Other Names: MT plus IS
  Arms: Medical treatment plus intracranial stenting (MT plus IS)
Drug: Medical treatment alone — This group will be given medical treatment including aspirin 100 mg and clopidogrel 75 mg per day for 90 consecutive days and clopidogrel 75 mg per day thereafter.
  Other Names: MT
  Arms: Medical treatment alone (MT)

SUMMARY:
In non-acute symptomatic ischemic stroke, the decision-making of medical treatment plus intracranial stenting has been more and more popular, especially in patients with intracranial large severe stenosis or occlusive artery. Nonetheless, there is no evidence from randomized controlled trials evaluating the efficacy of this treatment after the Wingspan Stent System Post Market Surveillance (WEAVE) and Wingspan One Year Vascular Imaging Events and Neurologic Outcomes (WOVEN) trial compared with medical treatment alone. This trial was to investigate whether medical treatment plus intracranial stenting would prevent the recurrent ischemic stroke in the territory of the symptomatic intracranial artery during 1-year follow-up.

DETAILED DESCRIPTION:
In symptomatic ischemic stroke due to intracranial large severe stenosis or occlusive artery, the choice for treatment has remained controversial after results of the Stenting versus Aggressive Medical Therapy for Intracranial Arterial Stenosis (SAMMPRIS) trial because it demonstrated that the efficacy of medical treatment was superior to intracranial stenting in the low risk of periprocedural stroke or death. However, this conclusion has influenced the role of intracranial stenting in the ischemic stroke treatment and recovery time for a long time because of the unproper patient selection of this trial such as no evidence of medical failure, intracranial stenting earlier than 7 days after the stroke and intracranial stenting in patients with transient ischemic attacks only. Recently, the Food and Drug Administration (FDA) mandated study about intracranial stenting, WEAVE trial, reported not only 97.4% patients with no complication at 72 hours, but also a relatively low 8.5% recurrent stroke and death rate during 1 year in the WOVEN study. In case of the symptomatic stenosis greater than 70%, the probability of recurrent stroke and transient ischemic attack in the territory of the symptomatic stenotic artery in 1 year was 23% and 14%, respectively, despite treatment with antithrombotic therapy and standard management of vascular risk. Given a lot of patients with symptomatic ischemic stroke who have some adjustable indications for intracranial stenting deployment in the world and a paucity of evidence from randomized trials, the purpose of this trial was to compare this treatment versus medical one in the intracranial large severe stenosis or occlusive artery.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of intracranial large severe stenosis or occlusive artery in angiography.
* Absence of intracranial hemorrhage.
* Premorbid mRS score is ≤ 3.
* Recurrent stroke in the target territory during the medical treatment for ischemic stroke prevention.

Exclusion Criteria:

* Tandem lesion.
* Loss to follow-up after discharge.
* A severe or fatal combined illness before acute ischemic stroke.
* Progressive neurologic deficit within 7 days after acute ischemic stroke.
* Large middle cerebral artery infarct within 30 days after acute ischemic stroke.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-05-24 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrent ischemic stroke of the qualifying lesion in the territory of the symptomatic intracranial artery. | During 1 year after randomization.
  Rate of recurrent ischemic stroke of the qualifying lesion in the territory of the symptomatic intracranial artery.

SECONDARY OUTCOMES:
Death rate of the qualifying lesion in the territory of the symptomatic intracranial artery. | During 1 year after randomization.
  Death rate of the qualifying lesion in the territory of the symptomatic intracranial artery.
Rate of ischemic stroke recovery of the qualifying lesion in the territory of the symptomatic intracranial artery. | During 3 months after randomization..
  Rate of ischemic stroke recovery of the qualifying lesion in the territory of the symptomatic intracranial artery was accessed by modified Rankin Score (mRS).

CONTACTS AND LOCATIONS:
Overall Officials: Cuong Tran Chi, Doctor, Study Chair — Can Tho SIS Hospital
Locations (1):
- Can Tho SIS Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Background] Alexander MJ, Zauner A, Chaloupka JC, Baxter B, Callison RC, Gupta R, Song SS, Yu W; WEAVE Trial Sites and Interventionalists. WEAVE Trial: Final Results in 152 On-Label Patients. Stroke. 2019 Apr;50(4):889-894. doi: 10.1161/STROKEAHA.118.023996. PMID 31125298
- [Background] Alexander MJ, Zauner A, Gupta R, Alshekhlee A, Fraser JF, Toth G, Given C, Mackenzie L, Kott B, Hassan AE, Shownkeen H, Baxter BW, Callison RC, Yu W. The WOVEN trial: Wingspan One-year Vascular Events and Neurologic Outcomes. J Neurointerv Surg. 2021 Apr;13(4):307-310. doi: 10.1136/neurintsurg-2020-016208. Epub 2020 Jun 19. PMID 32561658
- [Background] Zaidat OO, Fitzsimmons BF, Woodward BK, Wang Z, Killer-Oberpfalzer M, Wakhloo A, Gupta R, Kirshner H, Megerian JT, Lesko J, Pitzer P, Ramos J, Castonguay AC, Barnwell S, Smith WS, Gress DR; VISSIT Trial Investigators. Effect of a balloon-expandable intracranial stent vs medical therapy on risk of stroke in patients with symptomatic intracranial stenosis: the VISSIT randomized clinical trial. JAMA. 2015 Mar 24-31;313(12):1240-8. doi: 10.1001/jama.2015.1693. PMID 25803346
- [Background] Markus HS, Larsson SC, Dennis J, Kuker W, Schulz UG, Ford I, Clifton A, Rothwell PM. Vertebral artery stenting to prevent recurrent stroke in symptomatic vertebral artery stenosis: the VIST RCT. Health Technol Assess. 2019 Aug;23(41):1-30. doi: 10.3310/hta23410. PMID 31422789